CLINICAL TRIAL: NCT03313505
Title: PROtein S100B for Mild Trauma of the HEad in Emergency Patients
Acronym: PROMETHEE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Responsible Party: Sponsor
Other Study IDs: 16-09; 2016-A00901-50 (Other: ANSM)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who had been tested for S100B protein
  Interventions: Biological: S100B protein dosage
- Patients who have benefited from another strategy
  Interventions: Other: Brain CT scan

INTERVENTIONS:
Biological: S100B protein dosage — S100B protein dosage will be carried out, by a blood sample, on the earliest after admission and before 3th hour following brain injury S100B protein dosage will be left to the assessment of the emergency physician in charge of the patient
  Groups: Patients who had been tested for S100B protein
Other: Brain CT scan — No injected brain CT-scan, regardless of the time between the brain injury and the arrival in the emergency unit. Realization of CT-scan will be left to the assessment of the emergency physician in charge of the patient
  Groups: Patients who have benefited from another strategy

SUMMARY:
Brain injury is a frequent purpose for consultation in emergency services. Management of brain injury is time and resource consuming, combining clinical monitoring and imaging.

The stage prior to the management of the victims of brain injury is stratification of the severity, potential or proven.

Severe brain injury requires emergent brain CT-scan, ideally within one hour of the first medical contact. Patients requiring this strategy present with focused neurological deficit, Glasgow score <15 to 2 hours after the trauma, suspicion of open fracture of the skull or dish pan fracture, any signs of fracture of the skull base (hemotympanum, bilateral peri-orbital ecchymosis), otorrhea or rhinorrhea of cerebrospinal fluid, more than one episode of vomiting in adults, and posttraumatic convulsion. Patients benefiting from anticoagulant therapy are included in this category.

Victims of brain injury that do not fall into this category are considered less critical.

By definition, mild traumatic brain injury :

* a trauma of the cephalic extremity :
* whose Glasgow score (30 min after the trauma or during the consultation) is 13-15,
* associated with one or more of the following: confusion; disorientation; loss of consciousness of 30 min or less; post-traumatic amnesia of less than 24 hours; other transient neurological abnormalities (focal signs, epileptic seizures, non-surgical intracranial lesion).

Among these patients, some are considered at risk of developing intracerebral lesions. Nevertheless, it should be noted that the prevalence of hemorrhagic complications is radically different between patients with a Glasgow score of 13 and those with a score of 15. Thus, the recommendations suggest a brain scan without injection of contrast media within 4 to 8 hours for patients with the following characteristics :

* a retrograde amnesia of more than 30 minutes,
* a loss of consciousness or amnesia associated with:

  * either a risk mechanism (pedestrian overturned by a motor vehicle, ejection of a vehicle, falling by more than one meter),
  * or an age> 65 years,
  * or coagulation disorders, including the use of platelet aggregation therapy. Patients who fall outside this definition are considered low risk of complication and should not benefit of imaging.

Data from the scientific literature show that an early brain CT-scan allows identification of post-traumatic lesions in this population. Nevertheless, organizational problems, including the availability of the imaging, radiation, and disruption of surveillance related to patient displacement, are limitations to this strategy. In contrast, the low cost-effectiveness of CT scan is often advocated in patients with mild traumatic brain injury. For example, in the Octopus study, 52 of 1316 patients who received CT scan after mild head trauma had an intracerebral lesion. Among these patients, 39 (3%) had intracerebral lesion related to trauma; for 13 (1%) patients, the link with the trauma was uncertain.

In fact, the search of alternatives for a safer, more conservative, more efficient practice, one of the objectives of which is to limit the undue use of cerebral scanning. Thus, many teams have been interested in the use of biological variables to guide the decision to use imagery.

Among candidate biomarkers, the S100B protein has been the subject of many evaluations which allow it to be used in current practice. Indeed, the increase of the S100B protein carried out within 3 hours following a mild head trauma makes it possible to identify the patients at risk of intracerebral lesion and to target the indications of imaging.

The purpose of the registry is to describe the use, interpretation and performance of the S100B protein in its use at bedside in emergency medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Victims of mild head trauma at risk of complication :

  o Adult patients with head trauma with:
* retrograde amnesia of more than 30 minutes, or
* loss of consciousness or amnesia of the facts associated with:

  * Either a risky mechanism (pedestrian overturned by a motor vehicle, ejection of a vehicle, drop of more than one meter),
  * either An age> 65 years,
  * Either clotting disorders, including platelet aggregation therapy.
  * either Glasgow Score to 15
* Admitted to the emergency department within three hours of the traumatic event.

Exclusion Criteria:

* Refusal to participate at the study
* Patients with obstacle to 7 days follow up
* Pregnant women
* Patients not subject to an health insurance scheme in France or Monaco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the emergency unit with mild brain injury and meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 787 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluation of the number of brain CT-scan saved in patients who have been tested for S100B protein | 53 weeks
  Percentage (%)

SECONDARY OUTCOMES:
Comparison of supported patients with S100B protein assay or without S100B protein assay | 53 weeks
  Percentage (%)
Intensive treatment comparison of the patients included in the centers that carried out an "intensive implementation" of the use of the S100B protein and those included in the centers that provided the S100B protein | 53 weeks
  Percentage (%)
Quantification and evaluation of deviations to the algorithm | 53 weeks
  Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick CLAESSENS, PU-PH, Study Director — Centre Hospitalier Princesse Grace; Karim TAZAROURTE, PU-PH, Study Director — Hospices Civils de Lyon
Locations (15):
- France (14):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - AP-HP Centre Hospitalier Universitaire Henri-Mondor, Créteil
  - Hospices Civils de Lyon - Pôle Est, Lyon
  - AP-HM La Timone, Marseille
  - Centre Hospitalier de Metz-Thionville, Metz
  - Centre Hospitalier Universitaire de Nice, Hôpital Pasteur, Nice
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Carémeau, Nîmes
  - AP-HP Nord Lariboisière, Paris
  - AP-HP Sud Pitié-Salpêtrière, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Charles Nicolle, Rouen
  - CHU de Strasbourg, Strasbourg
  - HIA Sainte Anne, Toulon
  - Centre Hospitalier Universitaire de Toulouse - Hôpital Purpan, Toulouse
- Centre Hospitalier Princesse Grace, Monaco, Monaco